CLINICAL TRIAL: NCT00322387
Title: Treatment With Plerixafor in Multiple Myeloma or Non-Hodgkin's Lymphoma Patients to Increase the Number of Peripheral Blood Stem Cells When Given With A Mobilizing Regimen of Chemotherapy and G-CSF
Brief Title: Mobilization of Stem Cells With Plerixafor, Chemotherapy and G-CSF in Multiple Myeloma or Non-Hodgkin's Lymphoma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMD3100-2104
Record Dates: First submitted 2006-05-04; First posted 2006-05-05 (Estimated); Results first posted 2010-07-14 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-02

CONDITIONS: Lymphoma, Non-Hodgkin; Multiple Myeloma
Keywords: Non-Hodgkin's Lymphoma; Multiple Myeloma; Stem cell mobilization
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Multiple Myeloma | interventions — Granulocyte Colony-Stimulating Factor; plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Plerixafor PM (Experimental): Participants received chemotherapy and G-CSF mobilization for 7 days according to standard procedures at the study center. When participants achieved a target CD34+ count of ≥20 cells/µL, apheresis began. G-CSF was given daily in the morning on the days of apheresis. After the first apheresis, plerixafor (240 µg/kg) was administered each evening (approximately 10pm) followed by apheresis 10 to 11 hours later for up to 4 consecutive days.
  Called 'Cohort A' in protocol, study report and publications.
  Interventions: Drug: G-CSF and plerixafor
- Plerixafor AM (Experimental): Participants received chemotherapy and G-CSF mobilization for 7 days according to standard procedures at the study center. When participants achieved a target CD34+ count of ≥20 cells/µL, apheresis began. G-CSF was given daily in the morning on the days of apheresis. The morning of the second day after the first apheresis, plerixafor (240 µg/kg) was administered followed by apheresis 6 hours later. Plerixafor (240 µg/kg) was administered in the morning followed by apheresis 6 hours later for up to 4 consecutive days.
  Called 'Cohort B' in protocol, study report and publications.
  Interventions: Drug: G-CSF and plerixafor
- Low CD34+ Count/ Plerixafor PM (Experimental): Participants received chemotherapy and G-CSF mobilization for 7 days according to standard procedures at the study center. If participants had a CD34+ count of >=10 cells/µL but <20 cells/µL on 2 consecutive days, plerixafor (240 µg/kg) was given in the evening. G-CSF was administered and apheresis performed in the morning. Plerixafor (240 µg/kg) administered in the evening followed by G-CSF and apheresis 10 to 11 hours later was repeated for up to 4 consecutive days.
  Called 'Cohort C' in protocol, study report and publications.
  Interventions: Drug: G-CSF and plerixafor
- Plerixafor After Chemo (Experimental): This investigational cohort evaluated the effect of administering plerixafor before white blood cell recovery.
  Participants received mobilizing chemotherapy, followed by 5 consecutive days of G-CSF (10 µg/kg). Starting on the sixth day, participants received G-CSF (10 µg/kg) plus plerixafor (240 µg/kg) daily for up to 3 consecutive days. If CD34+ counts reached >= 20 cells/µL 6 hours after any of the 3 plerixafor doses, apheresis began. If not, G-CSF administration continued until the participant qualified for one of the other treatment arms.
  Called 'Investigational Cohort' in protocol, study report and publications.
  Interventions: Drug: G-CSF and plerixafor

INTERVENTIONS:
Drug: G-CSF and plerixafor — G-CSF and plerixafor were administered as described in the treatment arms.
  Other Names: Mozobil; AMD3100

SUMMARY:
Patients with multiple myeloma (MM) and non-Hodgkin's lymphoma (NHL) will be mobilized with chemotherapy and G-CSF plus plerixafor (AMD3100). The purpose of this protocol is to determine if plerixafor given after chemotherapy and G-CSF mobilization regimen is safe, if it can increase the circulating levels of peripheral blood stem cells (PBSCs) by ≥ 2-fold before apheresis, and if transplantation with the apheresis product was successful, as measured by time to engraftment of polymorphonuclear leukocytes (PMNs) and platelets (PLTs).

DETAILED DESCRIPTION:
An open label, multi-center, phase 2 study was conducted in patients with MM or NHL who were to be treated with peripheral blood stem cells (PBSC) autologous transplantation. The only change to the standard of care was the addition of plerixafor to a mobilization regimen of chemotherapy and G-CSF. Patients were first given a mobilizing regimen of chemotherapy as per local practice guidelines and G-CSF (at customary doses) and apheresis was performed. After the first apheresis, plerixafor was given at 10PM, 10-11 hours before the second apheresis the next day or in the morning of the second day, 6 hours before the second apheresis. The change in the patient's peripheral CD34+ cell count between the plerixafor dose and the start of apheresis was measured. The apheresis yields on Day 1 and Day 2 were compared.

This study was previously posted by AnorMED, Inc. In November 2006, AnorMED, Inc. was acquired by Genzyme Corporation. Genzyme Corporation is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria (Abbreviated List):

* MM in first partial response/complete response, first relapse, or second partial/complete response
* NHL in first or second partial or complete remission
* NHL patients who do not have bone marrow involvement and < 10% for follicular involvement
* MM patients who have stable disease with < 40% bone marrow involvement
* No more than three prior regimens of chemotherapy (thalidomide and Decadron are not considered chemotherapy)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* White blood cell count (WBC) >3.0 x 10^9/L
* Absolute neutrophil count >1.5 x 10^9/L
* Platelet count >100 x 10^9/L

Exclusion Criteria (Abbreviated List):

* Brain metastases or carcinomatous meningitis
* Hypercalcaemia [>1 mg/dl above the upper limit of normal (ULN)]
* Cardiovascular disease that includes proven or predisposition to ventricular arrhythmias
* Acute Infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-04; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (5):
- United States (5):
  - City of Hope National Medical Center, Duarte, California
  - Indiana Blood and Marrow Transplantation, Beech Grove, Indiana
  - University of Rochester Medical Center, Rochester, New York
  - Oregon Health and Science University, Portland, Oregon
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Result] Dugan MJ, Maziarz RT, Bensinger WI, Nademanee A, Liesveld J, Badel K, Dehner C, Gibney C, Bridger G, Calandra G. Safety and preliminary efficacy of plerixafor (Mozobil) in combination with chemotherapy and G-CSF: an open-label, multicenter, exploratory trial in patients with multiple myeloma and non-Hodgkin's lymphoma undergoing stem cell mobilization. Bone Marrow Transplant. 2010 Jan;45(1):39-47. doi: 10.1038/bmt.2009.119. Epub 2009 Jun 1. PMID 19483760

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with NHL or MM eligible for the study were recruited from 5 centers in the United States. The first patient was enrolled (signed informed consent) in April 2004 and the last patient's last study visit was July 2006.
Pre-assignment Details: Forty-four participants were enrolled; four participants never received plerixafor treatment so are excluded from summary tables.
Groups:
- Non-Hodgkin's Lymphoma (NHL): Participants with non-Hodgkin's lymphoma were assigned to Plerixafor PM, Plerixafor AM, and Plerixafor After Chemo treatment arms.
- Multiple Myeloma (MM): Participants with multiple myeloma were assigned to any of the 4 treatment arms.
Period: Treatment Period
Arm/Group | Non-Hodgkin's Lymphoma (NHL) | Multiple Myeloma (MM)
Started | 14 (Plerixafor PM=7, Plerixafor AM=6, Low CD34+ Count/Plerixafor PM=0, and Plerixafor After Chemo=1) | 26 (Plerixafor PM=12, Plerixafor AM=9, Low CD34+ Count/Plerixafor PM=1, and Plerixafor After Chemo=4)
Completed | 14 (Completed refers to completed all treatment visits.) | 25 (Completed refers to completed all treatment visits.)
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Follow-up Period
Arm/Group | Non-Hodgkin's Lymphoma (NHL) | Multiple Myeloma (MM)
Started | 14 (Participants who had transplants) | 26 (Participants who had transplants. One participant did not complete therapy but had a transplant.)
Completed | 12 (Follow-up visit 12 months post-transplant) | 23 (Follow-up visit 12 months post-transplant)
Not Completed | 2 | 3
Not completed — Final assessment not done | 1 | 3
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-Hodgkin's Lymphoma (NHL) | Multiple Myeloma (MM) | Total
Number analyzed (Participants) | 14 | 26 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (10.8) | 56.1 (7.6) | 55.6 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 6 | 15 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 14 | 24 | 38
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Participant Counts of Adverse Events (AEs) Up to Twelve Months Post Transplant
Description: Safety assessment was based on the incidence of adverse event reports. Participant count of AEs (Adverse Events) by severity and by relationship to study drug. AEs were reported regardless of relationship to study treatment. The investigator graded each AE using the World Health Organization (WHO) Adverse Event Grading Scale and provided assessments of seriousness and relatedness to study treatment.
Time Frame: 13 months
Population: Safety population who received at least one dose of plerixafor.
Measure: Number; unit: participants
Groups:
- Non-Hodgkin's Lymphoma (NHL): Plerixafor PM: Participants with NHL who followed the Plerixafor PM treatment arm regimen. Participants received chemotherapy and G-CSF mobilization for 7 days according to standard procedures at the study center. When participants achieved a target CD34+ count of ≥20 cells/µL, apheresis began. G-CSF was given daily in the morning on the days of apheresis. After the first apheresis, plerixafor (240 µg/kg) was administered each evening (approximately 10pm) followed by apheresis 10 to 11 hours later for up to 4 consecutive days.
- Non-Hodgkin's Lymphoma (NHL): Plerixafor AM: Participants with NHL who followed the Plerixafor AM treatment arm regimen. Participants received chemotherapy and G-CSF mobilization for 7 days according to standard procedures at the study center. When participants achieved a target CD34+ count of ≥20 cells/µL, apheresis began. G-CSF was given daily in the morning on the days of apheresis. The morning of the second day after the first apheresis, plerixafor (240 µg/kg) was administered followed by apheresis 6 hours later. Plerixafor (240 µg/kg) was administered in the morning followed by apheresis 6 hours later for up to 4 consecutive days.
- Non-Hodgkin's Lymphoma (NHL): Plerixafor After Chemo: Participants with NHL who followed the Plerixafor After Chemo treatment arm regimen. This investigational cohort evaluated the effect of administering plerixafor before white blood cell recovery.
  Participants received mobilizing chemotherapy, followed by 5 consecutive days of G-CSF (10 µg/kg). Starting on the sixth day, participants received G-CSF (10 µg/kg) plus plerixafor (240 µg/kg) daily for up to 3 consecutive days. If CD34+ counts reached >= 20 cells/µL 6 hours after any of the 3 plerixafor doses, apheresis began. If not, G-CSF administration continued until the participant qualified for one of the other treatment arms.
- Multiple Myeloma (MM): Plerixafor PM: Participants with MM who followed the Plerixafor PM treatment arm regimen. Participants received chemotherapy and G-CSF mobilization for 7 days according to standard procedures at the study center. When participants achieved a target CD34+ count of ≥20 cells/µL, apheresis began. G-CSF was given daily in the morning on the days of apheresis. After the first apheresis, plerixafor (240 µg/kg) was administered each evening (approximately 10pm) followed by apheresis 10 to 11 hours later for up to 4 consecutive days.
- Multiple Myeloma (MM): Plerixafor AM: Participants with MM who followed the Plerixafor AM treatment arm regimen. Participants received chemotherapy and G-CSF mobilization for 7 days according to standard procedures at the study center. When participants achieved a target CD34+ count of ≥20 cells/µL, apheresis began. G-CSF was given daily in the morning on the days of apheresis. The morning of the second day after the first apheresis, plerixafor (240 µg/kg) was administered followed by apheresis 6 hours later. Plerixafor (240 µg/kg) was administered in the morning followed by apheresis 6 hours later for up to 4 consecutive days.
- Multiple Myeloma (MM): Low CD34+ Count/Plerixafor PM: Participants with MM who followed the Low CD34+ Count/Plerixafor PM treatment arm regimen. Participants received chemotherapy and G-CSF mobilization for 7 days according to standard procedures at the study center. If participants had a CD34+ count of >=10 cells/µL but <20 cells/µL on 2 consecutive days, plerixafor (240 µg/kg) was given in the evening. G-CSF was administered and apheresis performed in the morning. Plerixafor (240 µg/kg) administered in the evening followed by G-CSF and apheresis 10 to 11 hours later was repeated for up to 4 consecutive days.
- Multiple Myeloma (MM): Plerixafor After Chemo: Participants with MM who followed the Plerixafor After Chemo treatment arm regimen. This investigational cohort evaluated the effect of administering plerixafor before white blood cell recovery.
  Participants received mobilizing chemotherapy, followed by 5 consecutive days of G-CSF (10 µg/kg). Starting on the sixth day, participants received G-CSF (10 µg/kg) plus plerixafor (240 µg/kg) daily for up to 3 consecutive days. If CD34+ counts reached >= 20 cells/µL 6 hours after any of the 3 plerixafor doses, apheresis began. If not, G-CSF administration continued until the participant qualified for one of the other treatment arms.
Arm/Group | Non-Hodgkin's Lymphoma (NHL): Plerixafor PM | Non-Hodgkin's Lymphoma (NHL): Plerixafor AM | Non-Hodgkin's Lymphoma (NHL): Plerixafor After Chemo | Multiple Myeloma (MM): Plerixafor PM | Multiple Myeloma (MM): Plerixafor AM | Multiple Myeloma (MM): Low CD34+ Count/Plerixafor PM | Multiple Myeloma (MM): Plerixafor After Chemo | All Participants
Number analyzed (Participants) | 7 | 6 | 1 | 12 | 9 | 1 | 4 | 40
participants
  Participants reporting ≥ 1 Adverse Event | 7 | 6 | 1 | 12 | 9 | 1 | 3 | 39
  AE Severity (Mild) | 3 | 3 | 0 | 2 | 2 | 0 | 0 | 10
  AE Severity (Moderate) | 2 | 1 | 1 | 6 | 3 | 0 | 2 | 15
  AE Severity (Severe) | 2 | 2 | 0 | 4 | 4 | 1 | 1 | 14
  AE Severity (Life Threatening) | 1 | 1 | 0 | 2 | 3 | 0 | 0 | 7
  AE Relationship to Drug (Not related) | 0 | 5 | 0 | 0 | 2 | 0 | 2 | 9
  AE Relationship to Drug (Probably not related) | 3 | 0 | 0 | 3 | 0 | 0 | 0 | 6
  AE Relationship to Drug (Possibly related) | 1 | 0 | 0 | 3 | 5 | 0 | 0 | 9
  AE Relationship to Drug (Probably related) | 1 | 1 | 1 | 3 | 1 | 0 | 0 | 7
  AE Relationship to Drug (Definitely related) | 2 | 0 | 0 | 3 | 1 | 1 | 1 | 8

2. Secondary Outcome: Fold (i.e., Relative) Increase in Peripheral Blood (PB) CD34+ Cells/µL
Description: The fold increase was measured by fluorescence activated cell sorting (FACS) analysis and was expressed as a ratio. Fold increase = (pre-apheresis PB CD34+ cells/µL)/(pre-plerixafor dosing PB CD34+ cells/µL).
Time Frame: Days 4-5 (first dose of plerixafor to apheresis)
Population: Intent to treat population. One participant in the Non-Hodgkin's Lymphoma (NHL): Plerixafor AM treatment group and 3 participants in the Multiple Myeloma (MM): Plerixafor After Chemo treatment group did not have samples taken for PB CD34+ cell counts on Day 1 and therefore could not be included.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Non-Hodgkin's Lymphoma (NHL): Plerixafor PM | Non-Hodgkin's Lymphoma (NHL): Plerixafor AM | Non-Hodgkin's Lymphoma (NHL): Plerixafor After Chemo | Multiple Myeloma (MM): Plerixafor PM | Multiple Myeloma (MM): Plerixafor AM | Multiple Myeloma (MM): Low CD34+ Count/Plerixafor PM | Multiple Myeloma (MM): Plerixafor After Chemo
Number analyzed (Participants) | 7 | 5 | 1 | 12 | 9 | 1 | 1
ratio | 2.2 (0.8) | 1.5 (0.8) | 1.2 (0.0) | 1.8 (0.4) | 6.5 (14.7) | 24.0 (0.0) | 3.1 (0.0)

3. Secondary Outcome: Number of Transplants in Which Participants Achieved Polymorphonuclear Leukocyte (PMN) Engraftment by Day 12 But No Later Than Day 21 Post Peripheral Blood Stem Cell (PBSC) Transplant
Description: Participants were monitored for polymorphonuclear leukocyte (PMN) engraftment as per the local standard of care. The target for engraftment was 12 days after PBSC transplant and no transplant taking longer than 21 days for engraftment.
Time Frame: 2 months
Population: Intent to treat population. Six participants with MM had 2 transplants.
Measure: Number; unit: transplants
Units Other Than Participants: transplants
Arm/Group | Non-Hodgkin's Lymphoma (NHL): Plerixafor PM | Non-Hodgkin's Lymphoma (NHL): Plerixafor AM | Non-Hodgkin's Lymphoma (NHL): Plerixafor After Chemo | Multiple Myeloma (MM): Plerixafor PM | Multiple Myeloma (MM): Plerixafor AM | Multiple Myeloma (MM): Low CD34+ Count/Plerixafor PM | Multiple Myeloma (MM): Plerixafor After Chemo
Number analyzed (Participants) | 7 | 6 | 1 | 12 | 9 | 1 | 4
Number analyzed (transplants) | 7 | 6 | 1 | 14 | 12 | 2 | 4
transplants
  ≤ Day 12 | 6 | 4 | 0 | 14 | 9 | 1 | 0
  Day 13 to Day 21 | 1 | 2 | 1 | 0 | 3 | 1 | 4
  ≥ Day 22 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment Period includes the first day of G-CSF mobilization to the day prior to chemotherapy/ablative treatment in preparation for the first transplant. This period includes G-CSF administration, the plerixafor dose, and the rest period.
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables. Each AE table includes events, regardless of reported relationship to study treatment or grade.
Groups:
- Non-Hodgkin's Lymphoma (NHL): Plerixafor After Chemo: Participants with NHL who followed the Plerixafor After Chemo treatment arm regimen.
  Participants received mobilizing chemotherapy, followed by 5 consecutive days of G-CSF (10 µg/kg). Starting on the sixth day, participants received G-CSF (10 µg/kg) plus plerixafor (240 µg/kg) daily for up to 3 consecutive days. If CD34+ counts reached >= 20 cells/µL 6 hours after any of the 3 plerixafor doses, apheresis began. If not, G-CSF administration continued until the participant qualified for one of the other treatment arms.
- Multiple Myeloma (MM): Low CD34+ Count/Plerixafor PM: Participants with MM who followed the Low CD34+ Count/Plerixafor PM treatment arm regimen.
  Participants received chemotherapy and G-CSF mobilization for 7 days according to standard procedures at the study center. If participants had a CD34+ count of >=10 cells/µL but <20 cells/µL on 2 consecutive days, plerixafor (240 µg/kg) was given in the evening. G-CSF was adminstered and apheresis performed in the morning. Plerixafor (240 µg/kg) administered in the evening followed by G-CSF and apheresis 10 to 11 hours later was repeated for up to 4 consecutive days.
- Multiple Myeloma (MM): Plerixafor After Chemo: Participants with MM who followed the Plerixafor After Chemo treatment arm regimen.
  Participants received mobilizing chemotherapy, followed by 5 consecutive days of G-CSF (10 µg/kg). Starting on the sixth day, participants received G-CSF (10 µg/kg) plus plerixafor (240 µg/kg) daily for up to 3 consecutive days. If CD34+ counts reached >= 20 cells/µL 6 hours after any of the 3 plerixafor doses, apheresis began. If not, G-CSF administration continued until the participant qualified for one of the other treatment arms.
Arm/Group | Non-Hodgkin's Lymphoma (NHL): Plerixafor PM | Non-Hodgkin's Lymphoma (NHL): Plerixafor AM | Non-Hodgkin's Lymphoma (NHL): Plerixafor After Chemo | Multiple Myeloma (MM): Plerixafor PM | Multiple Myeloma (MM): Plerixafor AM | Multiple Myeloma (MM): Low CD34+ Count/Plerixafor PM | Multiple Myeloma (MM): Plerixafor After Chemo
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/6 | 0/1 | 2/12 | 2/9 | 0/1 | 1/4
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6 | 1/1 | 12/12 | 9/9 | 1/1 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-Hodgkin's Lymphoma (NHL): Plerixafor PM (N=7) | Non-Hodgkin's Lymphoma (NHL): Plerixafor AM (N=6) | Non-Hodgkin's Lymphoma (NHL): Plerixafor After Chemo (N=1) | Multiple Myeloma (MM): Plerixafor PM (N=12) | Multiple Myeloma (MM): Plerixafor AM (N=9) | Multiple Myeloma (MM): Low CD34+ Count/Plerixafor PM (N=1) | Multiple Myeloma (MM): Plerixafor After Chemo (N=4)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 1 — Five participants experienced neutropenia starting before the first dose of plerixafor.
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 — One participant experienced stapylococcal sepsis immediately after salvage chemotherapy 24 days after the participant received plerixafor.
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-Hodgkin's Lymphoma (NHL): Plerixafor PM (N=7) | Non-Hodgkin's Lymphoma (NHL): Plerixafor AM (N=6) | Non-Hodgkin's Lymphoma (NHL): Plerixafor After Chemo (N=1) | Multiple Myeloma (MM): Plerixafor PM (N=12) | Multiple Myeloma (MM): Plerixafor AM (N=9) | Multiple Myeloma (MM): Low CD34+ Count/Plerixafor PM (N=1) | Multiple Myeloma (MM): Plerixafor After Chemo (N=4)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 6 | 3 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 0 | 0 | 6 | 7 | 0 | 1
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0
Rectal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0
Catheter related complication (General disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0
Catheter site discharge (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Catheter site erythema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Catheter site haemorrhage (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Catheter site pain (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Disease progression (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 2 | 1 | 0 | 0
Infusion site vesicles (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Injection site erythema (General disorders) | 2 | 0 | 0 | 2 | 1 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site pruritus (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site urticaria (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nail infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Carbon monoxide diffusing capacity decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 2 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 2 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0 | 7 | 7 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1 | 3 | 0 | 0
Headache (Nervous system disorders) | 5 | 0 | 1 | 2 | 3 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 3 | 2 | 1 | 3 | 1 | 0 | 0
Sensory loss (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 0
Nightmare (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Genital lesion (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Periorbital oedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The number and complexity of the cohorts make generalizations regarding the data problematic. Each cohort was small, and mobilizing and high-dose conditioning regimens varied across sites. AEs may include residual effects of chemotherapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after Genzyme publishes or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.